CLINICAL TRIAL: NCT04412785
Title: Phase I Trial for the Prevention of Cytokine Release Syndrome (CRS) With Cyclosporine in Patients With Moderate COVID-19
Brief Title: Cyclosporine in Patients With Moderate COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 842998
Record Dates: First submitted 2020-06-01; First posted 2020-06-02 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Cyclosporine; oral or IV route of administration, per investigator discretion. Duration of administration up to 14 days, as tolerated.
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine — • The initial dose will be 9 mg/kg/day oral divided q12h. For IV, the dose will be 3mg/kg/day by continuous IV infusion.
  Other Names: Sandimmune, Neoral, Gengraf

SUMMARY:
Phase 1 safety study to determine the tolerability, clinical effects, and changes in laboratory parameters of short course oral or IV cyclosporine (CSA) administration in patients with COVID-19 disease requiring oxygen supplementation but not requiring ventilator support.

DETAILED DESCRIPTION:
Our overall hypothesis is that CSA is safe in this patient population and that it will have antiviral and anti-cytokine effects as measured in laboratory tests.

The initial dose will be 9 mg/kg/day oral divided q12h or 3 mg/kg/day by continuous IV infusion. Oral administration is generally preferred, however IV administration can be used if oral administration is not feasible or cannot be tolerated, or at the physician-investigator's clinical discretion. The dose will be adjusted to target a trough level of 200 to 300 ng/ml, which is in alignment with common clinical practice. The planned duration of CSA treatment is up to 14 days, with planned discontinuation upon discharge from the hospital. Dose reduction of 25% to 50% can be made for patients who experience adverse events such as hypertension or serum creatinine elevation.

The end of study will be study day 30 for those patients who have been discharged from the hospital. If the patient remains in the hospital, the subject will still complete the end of study visit at day 30 as planned, but will continue to be followed until date of discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged >18.
4. Admitted to hospital with laboratory confirmation of SARS-CoV-2 infection.
5. Estimated creatinine clearance >50 ml/min using standard Cockcroft-Gault formula.

Exclusion Criteria:

1. Are admitted to the ICU at time of enrollment.
2. Have an active uncontrolled infection with a non-COVID-19 agent.
3. Have an active malignancy, not including non-melanoma skin cancer, superficial cervical or bladder cancer, MGUS, or prostate cancer with PSA <1.0.
4. Are on chronic immune suppressive medications, including
5. corticosteroid therapy at a prednisone equivalent dose of 10 mg per day or higher; therapy with calcineurin inhibitors or mTOR inhibitors.
6. Are pregnant
7. Are lactating
8. Have a known allergic reaction to components of the CSA or its diluents.
9. Are receiving investigational vaccine for SARS-CoV-2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Safety-oxygen, ICU transfer and ventilation | 3 months
  Safety will be measured: By assessing the proportion of participants requiring increase in oxygen requirements, transfer to intensive care unit, and/or mechanical ventilation
Safety-changes in absolute lymphocyte count | 3 months
  Safety will be assessed: By monitoring changes in absolute lymphocyte counts
Safety-changes in creatinine clearance | 3 months
  Safety will be assessed: By monitoring changes in creatinine clearance. Creatinine clearance will be estimated using the Cockcroft-Gault formula.
Safety-secondary bacterial infections | 3 months
  Safety will be assessed: By monitoring the incidence of secondary bacterial infections complicating COVID-19 hospitalization

SECONDARY OUTCOMES:
Laboratory measurements of safety and antiviral efficacy related to COVID-19-SARS-CoV-2 by measuring the clearance of SARS-CoV-2 from respiratory secretions | 3 months
  To measure time to SARS-CoV-2 clearance (PCR negativity) at Days 7 and 14 by deep nasal swab
Laboratory measurements-D-dimer levels | 3 months
  To measure the laboratory correlatives of CRS/ Hemophagocytic lymphohistiocytosis (HLH) by measuring: D-dimer levels
Laboratory measurements-ferritin | 3 months
  To measure the laboratory correlatives of CRS/ Hemophagocytic lymphohistiocytosis (HLH) by measuring: ferritin levels
Laboratory measurements- IL-6 | 3 months
  To measure the laboratory correlatives of CRS/ Hemophagocytic lymphohistiocytosis (HLH) by measuring: IL-6 levels

CONTACTS AND LOCATIONS:
Overall Officials: Emily Blumberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Blumberg EA, Noll JH, Tebas P, Fraietta JA, Frank I, Marshall A, Chew A, Veloso EA, Carulli A, Rogal W, Gaymon AL, Schmidt AH, Barnette T, Jurek R, Martins R, Hudson BM, Chavda K, Bailey CM, Church SE, Noorchashm H, Hwang WT, June CH, Hexner EO. A phase I trial of cyclosporine for hospitalized patients with COVID-19. JCI Insight. 2022 Jun 8;7(11):e155682. doi: 10.1172/jci.insight.155682. PMID 35536669